CLINICAL TRIAL: NCT04079517
Title: A Randomized, Open Pilot Study to Investigate the Mammographic Density Reduction on Healthy Women, Within the Karma Cohort, for Two Different Doses of Tamoxifen
Brief Title: Karolinska Interventional Study of Mammograhic Density (Karisma-1)
Acronym: Karisma-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Hall, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-000345; 2014-005005-20 (EudraCT Number)
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Mammographic Density
Keywords: Tamoxifen; Low-dose; Randomized Clinical Trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamoxifen 10mg (Experimental): Randomised dose of daily oral Tamoxifen 10mg, for 180 days
  Interventions: Drug: Tamoxifen
- Tamoxifen 20mg (Active Comparator): Randomised dose of daily oral Tamoxifen 20mg, for 180 days
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — A registered SERM drug, Tamoxifen.

SUMMARY:
A feasibility study, randomising to either 10 or 20 mg of tamoxifen. The primary aim is to identify the time to mammographic density change and piloting the procedures. It is known that a density change is seen after 12 months of 20 mg of tamoxifen, but the clinical experience indicates that an effect of drugs influencing mammographic density could be seen already after a few months. The second aim is to evaluate if there is a density change from 10 mg of tamoxifen equivalent to 20 mg.

DETAILED DESCRIPTION:
The investigators want to conduct a feasibility study including 42 women who will be randomised to either 10 or 20 mg of daily oral tamoxifen. The primary aim of the study is to identify the time to mammographic density change and piloting the procedures. It is known that a density change is seen after 12 months of 20 mg of daily tamoxifen, but the clinical experience indicates that an effect of drugs influencing mammographic density could be seen already after a few months. The second aim of the pilot study is to see if there is a density change from 10 mg of tamoxifen equivalent to 20 mg and if there is a difference in adverse reactions between the two doses. Interim analysis will be performed at 6 months, monitoring both safety and level of mammographic density change.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in the Karma study
* Attending the national mammography screening program, i.e. aged 40-74
* A mammogram, including a stored raw image, must have been taken within 3 weeks of baseline and start of therapy
* Having a mammographic volumetric density above the lowest 1/6, measured by Volpara
* Informed consent must be signed before any study specific assessments have been performed

Exclusion Criteria:

* Being pregnant or planning to become pregnant during the study
* Any previous or current diagnosis of breast cancer (including carcinoma in situ)
* Recalled (mammographic code 3 or above) after baseline screening mammography
* Any previous diagnosis of cancer, with the exception of non-melanoma skin cancer and in situ cancer of the cervix
* Currently using oestrogen and progesterone-based hormone replacement therapy
* Current use of hormone contraceptive with hormones, e.g. hormonal contraceptive pills, or progesterone implants. Hormonal intrauterine devices are accepted.
* A history of thromboembolic disease such as embolism, deep vein thrombosis, stroke, TIA or cardiac arrest.
* A history of immobilization, e.g. using wheelchair
* Uncontrolled diabetes defined as known untreated diabetes
* Hypertension at baseline, defined as systolic pressure higher than 140 mm Hg and diastolic higher than 90 mm Hg
* Use of drugs that interfere with CYP2D6 expression such as paroxetine, fluoxetine and bupropion

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hall, MD, PhD, Principal Investigator — Karolinska Institutet

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamoxifen 10mg | Tamoxifen 20mg
Started | 23 | 19
Completed | 18 | 15
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen 10mg | Tamoxifen 20mg | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.74 (8.48) | 62.32 (6.74) | 61.5 (5.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Breast Density
Description: Mean change in mammographic breast density at 6 months compared to baseline (=0 months) for each dose arm, using the fully automated STRATUS method. The average percent density (fibroglandular dense tissue area divided by total breast area) of left and right breasts at baseline was calculated and compared with average percent density at the end of the trial period and density change was defined as the difference between these two measures.
Time Frame: 6 months
Population: The final analysis was restricted to the 19 plus 14 participants.
Measure: Mean (95% Confidence Interval); unit: percentage of breast area
Groups:
- Tamoxifen 10mg: Randomised dose of daily oral Tamoxifen 10mg, for 270 days. Tamoxifen: A registered SERM drug, Tamoxifen.
- Tamoxifen 20mg: Randomised dose of daily oral Tamoxifen 20mg, for 270 days. Tamoxifen: A registered SERM drug, Tamoxifen.
Arm/Group | Tamoxifen 10mg | Tamoxifen 20mg
Number analyzed (Participants) | 19 | 14
percentage of breast area | -3.3 [-6.1 to -0.5] | -2.5 [-2.5 to 0.8]

2. Secondary Outcome: Symptom Score
Description: Symptom score change, compared to baseline for each dose arm. Questionnaires were used at 0, 1, 3, 6, 9 months. Vasomotor, gynecological, sexual, and musculoskeletal symptoms were assessed using a 5-grade Likert severity scale ranging from "no symptom at all" to "very much symptoms". A higher symptom score equals less symptoms, i.e. a better outcome.
  The questionnaire was based on the Functional Assessment of Cancer Therapy - Endocrine Subscale 7 (FACT-ES.7).
  The presented score was calculated as the sum of the last month's symptom severity levels and are presented as the absolute differences in symptom score on a scale ranging from any minus five to any plus five. A higher symptom score equals less symptoms, i.e. a better outcome.
Time Frame: 9 months
Population: Participants answering baseline and 9 month questionnaires.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tamoxifen 10mg | Tamoxifen 20mg
Number analyzed (Participants) | 18 | 12
score on a scale | 1.8 [-0.8 to 4.5] | 3.7 [0.5 to 6.8]
Statistical Analysis 1: Comparison: Tamoxifen 10mg vs Tamoxifen 20mg; Test type: Non-Inferiority — Comparing mean difference in symptom score (95% confidence intervals). Post hoc analysis. Not powered, but to give an indication of differences between standard dose (20mg) and the non-approved dose (10mg); Mean Difference (Final Values) = 1.9 — Post hoc analysis. Not powered, but to give an indication on differences in symptom score between standard dose (20mg) and the non-approved dose (10mg); Post hoc analysis. Not powered, but to give an indication on differences between standard dose (20mg) and the non-approved dose (10mg)

ADVERSE EVENTS:
Arm/Group | Tamoxifen 10mg | Tamoxifen 20mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 18/23 | 18/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen 10mg (N=23) | Tamoxifen 20mg (N=19)
Numbness/tingling in the hands and feet (Nervous system disorders) | 3 (3) | 5 (5)
Mood swings (Nervous system disorders) | 6 (6) | 6 (6)
Headaches (Nervous system disorders) | 10 (10) | 9 (9)
Concentration ability impaired (Nervous system disorders) | 1 (1) | 2 (2)
Feeling sad (Nervous system disorders) | 3 (3) | 5 (5)
Irritable (Nervous system disorders) | 5 (5) | 7 (7)
Lack of energy (Nervous system disorders) | 6 (6) | 7 (7)
Worry (Nervous system disorders) | 7 (7) | 6 (6)
Eyesight changes (Nervous system disorders) | 6 (6) | 8 (8)
Difficulty sleeping (Nervous system disorders) | 11 (11) | 9 (9)
Feel lightheaded (dizzy) (Nervous system disorders) | 4 (4) | 4 (4)
Vaginal bleeding or spotting (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 7 (7) | 11 (11)
Sexual feeling decreased (Reproductive system and breast disorders) | 9 (9) | 10 (10)
Vaginal itching/irritation (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Pain from breast tissue or breast skin (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Fragile mucous membranes/ Mucous membrane disorder (Reproductive system and breast disorders) | 7 (7) | 10 (10)
Painful intercourse (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Dryness vaginal (Reproductive system and breast disorders) | 11 (11) | 14 (14)
skin rashes (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Hair loss (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Problems with urination (Renal and urinary disorders) | 2 (2) | 3 (3)
Cold sweat (Endocrine disorders) | 8 (8) | 9 (9)
Night sweats (Endocrine disorders) | 15 (15) | 18 (18)
Menopausal hot flushes (Endocrine disorders) | 14 (14) | 17 (17)
muscle cramps (e.g. in legs) (Musculoskeletal and connective tissue disorders) | 14 (14) | 16 (16)
Pain in joints (Musculoskeletal and connective tissue disorders) | 12 (12) | 11 (11)
Diarrhoea (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Constipation (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
weight gain (Metabolism and nutrition disorders) | 12 (12) | 14 (14)
Nausea (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Vomiting (Metabolism and nutrition disorders) | 12 (12) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes